CLINICAL TRIAL: NCT04249921
Title: Evaluation of Acupuncture Effects for Complications After Surgery of Cerebellopontine Angle Tumor in Skull Base
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019-09-001AU
Record Dates: First submitted 2019-12-08; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Acupuncture; Tumor, Brain; Skull Base Tumor; Cerebellopontine Angle Tumor; Complication of Treatment; Quality of Life; Neuromuscular Blockade
MeSH Terms: conditions — Brain Neoplasms; Skull Base Neoplasms; Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: 1. Use acupuncture to treat the patients who received the surgery of CPA tumor. Acupoints of reference: Yifeng(TE17),Tinggong(SI19),Xiaguan(ST07),Wind Pool(GB20),Outer Pass(SJ5),Union Valley(LI4),Yang Mound Spring(GB34),Leg Three Li(ST36).
  2. Use questionnaires to evaluate.The questionnaires including House-Brackmann Grading Scale,WHOQOL-BREF Taiwan Version,Functional Assessment of Cancer Therapy: General(FACT-G),Visual Analogue Scale(VAS).
- Control: 1.Use questionnaires to evaluate.The questionnaires including House-Brackmann Grading Scale,WHOQOL-BREF Taiwan Version,Functional Assessment of Cancer Therapy: General(FACT-G),Visual Analogue Scale(VAS).

SUMMARY:
Skull base tumors are a type of tumor that grow in the area of several skulls behind the cranial cavity. The incidence rate is 2 to 18 per 100,000 people per year; males and females are likely to have a proportional difference in the types of skull base tumors.

Cerebellopontine angle (CPA) tumors are the most common neoplasms in the posterior skull base,accounting for 5-10% of skull base tumors.Some different kinds of tumors can grow in cerebellopontine angle. The tumors are more likely to cause some symptoms when they grow large enough to put pressure on the brain.

A common traditional treatment for skull base tumors is neurosurgery-craniotomy. However, after the operation, brain may be injured with hematoma, and the instruments used are in contact with the brain. It is still inevitable that there will have complications of minor and major nerve damages, such as facial paralysis,trigeminal neuralgia, tinnitus, sports disorders (ataxia) and so on.

Acupuncture has a unique effect on the treatment of the human nervous system. Aim of the study is used acupuncture to improve the complications of the surgery of Cerebellopontine angle tumors in skull base.

DETAILED DESCRIPTION:
Skull base has clinically unique importance:it is the anatomic junction of the neural and facial viscerocranium,supports human brain and supports that contains the neurovascular structures entering or exiting the skull,it divided into anterior,middle and posterior skull base.Skull base tumors are a type of tumor that grow in the area of several skulls behind the cranial cavity ,tumors most grow inside the skull base, and a few are formed outside because the tumor may originate from the base of skull or elsewhere in the body (metastatic).The incidence rate is 2 to 18 per 100,000 people per year; males and females are likely to have a proportional difference in the types of skull base tumors.

Cerebellopontine angle (CPA) tumors are common skull base tumors in posterior skull base. CP angle located below the cerebrum, between the pons and the cerebellum and between the superior and inferior limbs of the cerebellopontine fissure, it is a V-shaped angular cleft. About 6%-10% of skull base tumors are in the cerebellopontine angle (CPA). 90% of tumors in this area(CPA) are vestibular schwannoma (acoustic neuromas), 3% are meningioma, and the rest are primary cholesteatoma (lipoma),facial nerve schwannoma ,angioma as well as arachnoid cyst etc..

At present, computed tomography (CT) and nuclear magnetic resonance imaging (MRI) can be used to detect and evaluate skull base lesions. When these tumors grow enough to compress the nerves around the brain, the areas where the tumor are pressed could cause some symptoms such as blurred vision, headache, dizziness and other specific symptoms that affect normal life.

A common traditional treatment for skull base tumors is neurosurgery-craniotomy. However, after the operation, the brain may be injured with hematoma, and the instruments used are in contact with the brain. It is still inevitable that there will have complications of minor and major nerve damages, such as facial paralysis and trigeminal neuralgia, tinnitus, sports disorders (ataxia) and so on. If the damages are in serious situations, patients are also possible to be serious infected or in a vegetative state.

Acupuncture has a unique effect on the treatment of the human nervous system. Acupuncture mainly aims to improve the complications of the surgery of Cerebellopontine angle tumors in skull base by eliminating blood stasis, clearing meridians, and strengthening the body.The researchers' selections of acupoints are distributed in Large Intestine,Stomach Meridian,Small Intestine Meridian,Triple Energizer Meridian and Gallbladder Meridian in body.

In the past, some researchers used questionnaires for the quality of life of skull base tumor surgery, and also some researchers used questionnaires to evaluate the efficacy of acupuncture. The rationale of the study is to combine these three-the surgery of CP Angle tumor in skull base,acupuncture and questionnaires.Namely,the researchers use four questionnaires to evaluate the efficacy of acupuncture after surgery of Cerebellopontine Angle tumor in skull base.

ELIGIBILITY:
Inclusion Criteria:

1. The patients who have been diagnosed Cerebellopontine Angle Tumor by neurosurgeons.
2. The Patients who have been undergoned the surgery of tumor
3. Not receiving acupuncture for other diseases (needle stimulate for body ) or any rehabilitation treatment at the same time
4. Voluntary participation in this study

Exclusion Criteria:

1. Taking anticoagulant drugs or who have coagulopathy
2. Pregnant women, especially pregnant women with habitual abortion
3. Skin infections
4. Acupuncture phobia (this study has invasive treatment: acupuncture)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients of cerebellopontine angle (CPA) tumors in skull base.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-10-04 (Estimated); Study Completion 2020-10-04 (Estimated)

PRIMARY OUTCOMES:
WHOQOL-BREF Taiwan Version | 8 weeks
  Evaluate the quality of life after acupuncture treatment, use WHOQOL-BREF Taiwan Version questionnaire. Scale: 0~100, higher scores, better life quality. Counted by each time recording and using mode conversion to get final scale.
Visual Analogue Scale: VAS | 8 weeks
  measurement for pain,to assess the pain degree. Scale: 0~100 mm, higher scores, higher pain . Counted by each time recording.
Functional Assessment of Cancer Therapy: General(FACT-G) | 8 weeks
  Evaluate the quality of life for " the patients of CPA tumor in skull base " after acupuncture treatment,there are four parts,physiology,social and family, emotion,function.Scale: 0~100, higher scores, better life quality. Counted by each time recording and using mode conversion to get final scale.
House-Brackmann grading scale | 8 weeks
  measurement and evaluate the level for the patients of facial paralysis after surgery of CPA tumor in skull base.Measure the upwards and outwards movement situation of eyebrows and mouth. Each reference point scores 1 point for each 0.25 cm movement, up to a maximum of 1 cm. The scores are then added together, to give a number out of 8.After that, the scale of facial paralysis corresponding to the score was divided into five levels, with the first level being the mildest and the fifth level being the most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Ta-Peng Wu, MD/Master, Study Director — tpwu@vghtpe.gov.tw
Locations (1):
- Center for Traditional Medicine, Taipei VGH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Memari F, Hassannia F, Abtahi SH. Surgical Outcomes of Cerebellopontine angle Tumors in 50 Cases. Iran J Otorhinolaryngol. 2015 Jan;27(78):29-34. PMID 25745609
- [Result] Bonneville F, Savatovsky J, Chiras J. Imaging of cerebellopontine angle lesions: an update. Part 1: enhancing extra-axial lesions. Eur Radiol. 2007 Oct;17(10):2472-82. doi: 10.1007/s00330-007-0679-x. Epub 2007 Jun 12. PMID 17562049
- [Result] Kunimatsu A, Kunimatsu N. Skull Base Tumors and Tumor-Like Lesions: A Pictorial Review. Pol J Radiol. 2017 Jul 25;82:398-409. doi: 10.12659/PJR.901937. eCollection 2017. PMID 28811848
- [Result] Gil Z, Fliss DM. Quality of life in patients with skull base tumors: current status and future challenges. Skull Base. 2010 Jan;20(1):11-8. doi: 10.1055/s-0029-1242979. PMID 20592852
- [Result] Roser F, Dimostheni A, Elhammady MS, Recinos P, Rigante L. Response to: Phillips M. et al. "Safety of commercial airflight in patients with brain tumors: a case series". Journal of Neuro-Oncology (2018) 139:617-623. J Neurooncol. 2019 Apr;142(2):393-394. doi: 10.1007/s11060-018-03088-6. Epub 2019 Jan 21. No abstract available. PMID 30666464
- [Result] Witgert ME, Veramonti T, Hanna E. Instruments for estimation of health-related quality of life in patients with skull base neoplasms. Skull Base. 2010 Jan;20(1):5-10. doi: 10.1055/s-0029-1242978. PMID 20592851
- [Result] Biswas D, Marnane C, Mal R, Baldwin D. Benign extracranial nerve sheath tumors of the skull base: postoperative morbidity and management. Skull Base. 2008 Mar;18(2):99-106. doi: 10.1055/s-2007-991109. PMID 18769654
- [Result] Xu S, Wang L, Cooper E, Zhang M, Manheimer E, Berman B, Shen X, Lao L. Adverse events of acupuncture: a systematic review of case reports. Evid Based Complement Alternat Med. 2013;2013:581203. doi: 10.1155/2013/581203. Epub 2013 Mar 20. PMID 23573135
- [Result] Chung A, Bui L, Mills E. Adverse effects of acupuncture. Which are clinically significant? Can Fam Physician. 2003 Aug;49:985-9. PMID 12943357
- [Result] Chen MH, Chen MH, Huang JS. Cervical subdural empyema following acupuncture. J Clin Neurosci. 2004 Nov;11(8):909-11. doi: 10.1016/j.jocn.2004.02.011. PMID 15519876
- [Result] Giovagnoli AR. Quality of life in patients with stable disease after surgery, radiotherapy, and chemotherapy for malignant brain tumour. J Neurol Neurosurg Psychiatry. 1999 Sep;67(3):358-63. doi: 10.1136/jnnp.67.3.358. PMID 10449559
- [Result] Zhang R, Wu T, Wang R, Wang D, Liu Q. Compare the efficacy of acupuncture with drugs in the treatment of Bell's palsy: A systematic review and meta-analysis of RCTs. Medicine (Baltimore). 2019 May;98(19):e15566. doi: 10.1097/MD.0000000000015566. PMID 31083225
- [Result] Qiu WQ, Claunch J, Kong J, Nixon EE, Fang J, Li M, Vangel M, Hui KK. The effects of acupuncture on the brain networks for emotion and cognition: an observation of gender differences. Brain Res. 2010 Nov 29;1362:56-67. doi: 10.1016/j.brainres.2010.09.040. Epub 2010 Sep 17. PMID 20851113
- [Result] Kim YD, Park JH, Yang SH, Kim IS, Hong JT, Sung JH, Son BC, Lee SW. Pain assessment in brain tumor patients after elective craniotomy. Brain Tumor Res Treat. 2013 Apr;1(1):24-7. doi: 10.14791/btrt.2013.1.1.24. Epub 2013 Apr 30. PMID 24904885
- [Result] Xiao X, Zheng Q, Shi Y, Zhang L, Zhao L, Zhou S, Zhang W, Cao W, Liu Y, Li Y. Association of Patients' Characteristics with Acupuncture Treatment Outcomes in Treating Bell's Palsy: Results from a Randomised Controlled Trial. Evid Based Complement Alternat Med. 2019 Aug 15;2019:6073484. doi: 10.1155/2019/6073484. eCollection 2019. PMID 31511780